CLINICAL TRIAL: NCT05779826
Title: The Effect of Playing Dough on Children's Adaptation to Nebulizer Treatment Children 3-6 Years Old Child Service: Randomized Controlled Study
Brief Title: Use of Play Dough in Children Receiving Nebulizer Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/02-23
Record Dates: First submitted 2023-02-24; First posted 2023-03-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nursing Caries; Nebulizer Therapy
Keywords: Nebulizer Therapy; Child; Play Dough; Adherence to treatment; Nursing; Play
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Play Dough Group (Experimental): Play dough was played while receiving nebulizer therapy for the children in play dough group.
  Interventions: Other: Play dough
- Routine Treatment Group (No Intervention): Play dough was not used for the children in the routine treatment group. Routine nebulizer treatment was applied to this group.

INTERVENTIONS:
Other: Play dough — In the play dough group, play dough was used during the treatment of children receiving nebulizer therapy.
  Arms: Play Dough Group

SUMMARY:
The aim of this study is to present the results of the effect of playing with play dough on treatment compliance in children aged 3-6 years receiving nebulizer therapy. In the randomized controlled study, 80 children who were hospitalized in the pediatric ward of a public hospital and met the inclusion criteria were equally divided into 2 groups. Play dough was played while receiving nebulizer therapy for the children in group 1 (research group). Play dough was not used for the children in the 2nd group. The compliance of the children in the two groups to the treatment was evaluated with the Child's Adherence to Nebulizer Treatment Evaluation Form (CANTEF).

DETAILED DESCRIPTION:
Mask use is generally preferred in children receiving nebulizer therapy. Wearing a mask and the noise made by the nebulizer device cause fear and stress in the child, leading to maladaptive behaviors such as crying, shouting, and trying to remove the mask. The aim of this study is to distract the child who receives nebulizer treatment by playing play dough and to present the results regarding compliance with the treatment.

Methods: This study was conducted in a single-center randomized controlled design. The sample size of the study was calculated in the program of G*Power 3.1.9.2 (Heinrich Heine University Düsseldorf, Germany). The sample size was found to be 35 children for each group. The research was conducted with a total of 80 children. There were 40 children in each group (research and control group). This study was carried out in the pediatric service of a public hospital in Istanbul between October 2021 and February 2022.

Procedures: The participants were divided into groups, the area to be played with play dough was prepared, vital signs were collected, data were collected with CANTEF and all recordings were made by the 1st researcher. She has 3 years of experience as a first research nurse.

In this study, the following procedure was applied respectively. Parents of children aged 3-6 years who are hospitalized in the pediatric service and who will be treated with nebulizers and who meet the sampling criteria will be informed about the study, and verbal and written consent will be obtained. A face-to-face interview method will be used to determine the socio-demographic and clinical characteristics of the children in data collection, and the data will be recorded in the Sick Child Diagnosis Form (SCDF) by the researcher. In order to evaluate the compliance of the children to the nebulizer treatment, the vital signs and behaviors will be evaluated by the researcher and the data will be recorded in the Child's Adherence to the Nebulizer Treatment Evaluation Form. For the random assignment of children to groups, children with an odd number of patient protocol numbers will form the research group, and children with an even number will form the control group. For example, the child with the protocol number 278861 was included in the research group, and the child with the protocol number 236724 was included in the control group. In this study, all evaluations were made in the same way for the children in the research and control groups. SCDF was filled in by obtaining information from the mother or father in the research group. 5 minutes before the nebulizer treatment, an area was created to play with play dough, the child was brought to a sitting position, vital signs were taken, his behavior was evaluated and recorded in the CANTEF. Nebulizer treatment was started at the beginning of the treatment (0. min), vital signs and behaviors were evaluated and recorded in the CANTEF, 5 minutes after the beginning of the treatment, vital signs and behaviors were evaluated and recorded in the CANTEF, 10 minutes after the start of the treatment, vital signs and behaviors were evaluated and recorded in the CANTEF, at the end of the treatment (15. min), the nebulizer treatment was terminated, the game activity was finished, and the behaviors were evaluated and recorded in the CANTEF. In the control group, the same procedures were performed in the same way without playing the play dough.

Instruments: Data were collected with the Sick Child Diagnosis Form (CSDFF) and the Child's Adherence to Nebulizer Treatment Evaluation Form (CANTEF). The forms were developed by the researchers based on the literature. The Sick Child Diagnosis Form (SCDF) is prepared for the child's age, gender, nationality, school attendance, whether he or she has been given nebulizer treatment before, if so, his reactions, reason for applying to the emergency department, diagnosis, whether he has a chronic disease, behavioral disorder such as attention deficit and hyperactivity disorder or not. It is a form consisting of 11 questions, which includes information about whether there is a diagnosed disease for respiratory diseases and whether there is a drug that he constantly uses if these diseases exist. While the first four questions determine the socio-demographic data of the child, the other seven questions describe the clinical features. Child's Adherence to Nebulizer Treatment Evaluation Form was prepared by the researcher and consultant to evaluate the vital signs and behaviors of children 5 minutes before the treatment, at the beginning of the treatment, 5 minutes after the start of the treatment, 10 minutes after the start of the treatment, and at the end of the treatment. In the evaluation of vital signs, there are 5 criteria: radial pulse, temporal fever, respiratory rate, respiratory function and SPO2. There are 10 behavioral criteria in the evaluation section of the child's behavior. For each behavioral criterion, there are two options, "yes" and "no". The 9th behavioral criterion will be evaluated from the beginning of the treatment (0. min). The 10th behavioral criterion will be evaluated only for the children in the research group. In the study, console type pulse oximeter, temporal thermometer and surgical mask were used in the research and control groups. In the research group, play dough was used during the treatment of children receiving nebulizer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Parent's consent to participate in the study
* Stable clinical status
* The child's motor skills should be at a level to be able to play with play dough and should be developed according to his age,
* The child's ability to speak and understand Turkish.

Exclusion Criteria:

* Any physical or mental disability that prevents the child from playing with play dough
* The child has a behavior disorder or disease that causes maladaptive behavior

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Identifying the child's adherence with nebulizer therapy | Children's behavior and vital signs were evaluated 5 minutes before the treatment. evaluated for 15 minutes during treatment. Evaluation was done every 5 minutes.
  The child's behavior during nebulizer therapy was assessed using the Child's Nebulizer Treatment Compliance Evaluation Form. In this form, body temperature, pulse, respiratory rate, saturation, respiratory function, and behaviors were evaluated. When assessing behaviors, she is "irritable", "crying", "not allowing her vital signs to be taken", "very active, not sitting up", "wanting to go to her parent's lap", "yelling and screaming" ', 'not communicating with the researcher', 'removing the mask from his face' criteria were evaluated. The answers were evaluated as "yes" or "no". Children with a high rate of yes answers were considered non-adherent to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Aydoğmuş, MSc, Principal Investigator — Martyr Prof. Dr. İlhan Varank Sancaktepe Education and Research Hospital
Locations (1):
- Maltepe University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ari A. Drug delivery interfaces: A way to optimize inhalation therapy in spontaneously breathing children. World J Clin Pediatr. 2016 Aug 8;5(3):281-7. doi: 10.5409/wjcp.v5.i3.281. eCollection 2016 Aug 8. PMID 27610343
- [Background] Caleffi CC, Rocha PK, Anders JC, Souza AI, Burciaga VB, Serapiao Lda S. Contribution of structured therapeutic play in a nursing care model for hospitalised children. Rev Gaucha Enferm. 2016 Jun;37(2):e58131. doi: 10.1590/1983-1447.2016.02.58131. Epub 2016 May 31. English, Portuguese. PMID 27253598
- [Background] DiBlasi RM. Clinical Controversies in Aerosol Therapy for Infants and Children. Respir Care. 2015 Jun;60(6):894-914; discussion 914-6. doi: 10.4187/respcare.04137. PMID 26070582
- [Background] Goralski JL, Davis SD. Breathing easier: addressing the challenges of aerosolizing medications to infants and preschoolers. Respir Med. 2014 Aug;108(8):1069-74. doi: 10.1016/j.rmed.2014.06.004. Epub 2014 Jun 25. PMID 25012949
- [Background] Hoiseth M, Keitsch MM, Holm Hopperstad M. Interactions between caregivers and young children: exploring pedagogical tact in nebulizer treatment. Qual Health Res. 2014 Dec;24(12):1622-34. doi: 10.1177/1049732314549017. Epub 2014 Sep 5. PMID 25192760
- [Background] Koller D, Goldman RD. Distraction techniques for children undergoing procedures: a critical review of pediatric research. J Pediatr Nurs. 2012 Dec;27(6):652-81. doi: 10.1016/j.pedn.2011.08.001. Epub 2011 Oct 13. PMID 21925588
- [Background] Lima KY, Santos VE. [Play as a care strategy for children with cancer]. Rev Gaucha Enferm. 2015 Jun;36(2):76-81. doi: 10.1590/1983-1447.2015.02.51514. Portuguese. PMID 26334412
- [Background] Shinta Devi NLP, Nurhaeni N, Hayati H. Effect of Audiovisual Distraction on Distress and Oxygenation Status in Children Receiving Aerosol Therapy. Compr Child Adolesc Nurs. 2017;40(sup1):14-21. doi: 10.1080/24694193.2017.1386966. PMID 29166200
- [Background] Stewart MW. Therapeutic Play Intervention. J Perianesth Nurs. 2016 Oct;31(5):452-6. doi: 10.1016/j.jopan.2016.07.001. No abstract available. PMID 27667353
- [Background] Ari A. A path to successful patient outcomes through aerosol drug delivery to children: a narrative review. Ann Transl Med. 2021 Apr;9(7):593. doi: 10.21037/atm-20-1682. PMID 33987291
- See also: A Guide To Aerosol Delivery Devices for Respiratory Therapists. American Association for Respiratory Care — https://www.aarc.org/wp-content/uploads/2015/04/aerosol_guide_rt.pdf